CLINICAL TRIAL: NCT01144897
Title: PET Acetate for Docetaxel Response Assessment in Hormone-Refractory Prostate Cancer
Brief Title: PET Acetate for Castrate-Resistant Prostate Cancer on Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Vaena (Other)
Responsible Party: Sponsor-Investigator, Daniel Vaena, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201002720
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Castrate Resistant Prostate Cancer; Prostate Cancer
Keywords: Castrate resistant; Prostate cancer; Docetaxel; Taxotere; PET Acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET Acetate Imaging with Docetaxel (Experimental): PET-acetate as an intermediate endpoint in the assessment of response of patients undergoing docetaxel for hormone refractory prostate cancer (HRPC).
  Subjects will be treated with docetaxel, 75 mg/m2 every 21 days until disease progression or unacceptable toxicity occurs. Subjects will have two PET acetate scans - one prior to beginning chemotherapy and one approximately 8-9 weeks after chemotherapy has begun.
  Interventions: Radiation: PET Acetate scan; Drug: Carbon-11 labeled Acetate

INTERVENTIONS:
Radiation: PET Acetate scan — PET Acetate scans will be done to detect prostate cancer lesions.
Drug: Carbon-11 labeled Acetate — C-11 Acetate is a radiotracer used in PET scanning
  Other Names: C-11 Acetate; Acetate

SUMMARY:
One purpose of this research study is to examine if a special type of imaging test, a positron emission tomography (PET) scan using the radioactive material [C-11] acetate, will be helpful in detecting prostate cancer lesions in subjects with castrate-resistant prostate cancer (CRPC). This PET scan will be combined with a computed tomography (CT) scan taken during the same imaging session. The other purpose of the PET-CT scan using [C-11] acetate (PET Acetate Scan) is to assist in identifying who is responding to the treatment (docetaxel chemotherapy).

DETAILED DESCRIPTION:
The purpose of the current pilot clinical trial is to attempt to identify the safety and accuracy of PET-acetate imaging in the assessment of response of persons undergoing first-line docetaxel for CRPC. If successful, the current research could lead to the incorporation of PET-acetate into future study protocols where continuation of chemotherapy is based on early PET-acetate results, provided that effective second-line therapy options are available (which is an expectation for the near future, based on several ongoing and presented phase III trials).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written consent document.
2. Patients must have histologically documented adenocarcinoma of the prostate at any time in the past.
3. At the time of enrollment: Patients must have evidence of castrate resistant metastatic prostate cancer (patients with rising PSA only and no other radiographic evidence of metastatic prostate cancer are not eligible). In addition, progressive disease is required as per #5 below.
4. Two categories of eligible patients exist: Measurable disease with any level of serum prostate-specific antigen (PSA) OR Non-measurable disease (positive bone scan) with PSA equal or greater than 2 ng/ml

   Definition of Measurable Disease/Target Lesions - Any lesion >/= 1 cm on spiral computed tomography (CT) that is believed to represent metastatic prostate cancer and that can be accurately measured in at least one dimension (longest diameter). However, if the lesion is a lymph node, it needs to be equal or greater than 20 mm (longest diameter) based on CT scans or physical exam (palpable lymph nodes). Chest X-ray with clearly defined lung lesions surrounded by aerated lung or parenchymal lung lesions measured as 10 mm or greater with a spiral CT are also eligible.

   Definition of Non-measurable Disease/Non-target Lesions - Non-target lesions include all other lesions not included above, including bone lesions. Previously irradiated lesions should not be used for eligibility unless progression was documented after radiation therapy.
5. In order to be eligible, patients must have demonstrated evidence of progressive disease prior to enrollment. Progressive disease is defined as any one of the following:

   * Measurable Disease Progression: Objective evidence of increase 20% or more in the sum of the longest diameters (LD) of target lesions from the time of maximal regression after prior therapy; or the appearance of one or more new lesions.
   * Bone Scan Progression: Appearance of two or more new lesions on bone scan. If no prior bone scan exists, presence of 2 lesions is needed for eligibility.
   * PSA Progression: An elevated PSA (2 ng/mL or higher) which has risen serially on at least two occasions at least each 1 week apart. Note: If patient was on antiandrogens as last therapy, 6 weeks need to elapse after discontinuation of the antiandrogen. For prior ketoconazole, 4 weeks need to elapse. If the confirmatory PSA (#2) value is less than the first rising PSA value, then an additional rising PSA (#3) will be required to document progression. For the purposes of this study, the last PSA value recorded prior to the initiation of treatment will be considered the baseline PSA.
6. Progression despite standard androgen deprivation therapy.
7. At least 4 weeks since any systemic steroids (any dose; unless used chronically for another illness at equal or less than 10 mg of prednisone daily, or in conjunction with prior ketoconazole resulting in slow steroid taper) and any other hormonal therapy.
8. No prior cytotoxic chemotherapy for prostate cancer.
9. Four weeks or longer since major surgery and fully recovered.
10. Four weeks or longer since any prior radiation (including palliative) and fully recovered.
11. No prior strontium or samarium.
12. Concurrent bisphosphonate use is allowed. However, if patient has not previously been on bisphosphonate, first dose should only occur after the baseline positron emission tomography (PET) acetate scan has been obtained.
13. ECOG performance status: 0-2
14. Age ≥ 18
15. Required Initial Laboratory Values (within 14 days of registration):

ANC ≥1500/microL; Platelet count ≥ 100,000/microL; Creatinine ≤1.5 x upper limits of normal; Bilirubin ≤ 1.5 x upper limits of normal; AST and ALT ≤ 1.5 x upper limits of normal; PSA level requirements: see #4; Serum Testosterone ≤ 50 ng/ dL (for patients who have not had bilateral orchiectomy); Estimated glomerular filtration rate > 30 mL/min

Exclusion Criteria:

1. No known brain metastases (brain imaging MRI/CT is not required unless clinical symptoms).
2. No current congestive heart failure (New York Heart Association Class III or IV).
3. No serious or non-healing wound, ulcer or bone fracture.
4. No peripheral neuropathy ≥ grade 2.
5. Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies are not eligible.
6. Patients who received prior docetaxel for any reason are not eligible.
7. PC-Spes, Saw Palmetto, and St. John's Wort must be discontinued before registration. The discontinuation of other herbal medications and food supplements is strongly encouraged. Patients may continue on daily vitamins and calcium supplements.
8. No known allergy to acetate.
9. No severe claustrophobia
10. Concurrent use of statins is allowed on study but use should not have started 30 days prior to entry into the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Interpretation of PET Acetate scans | Time of enrollment up to one year
  Standardized uptake values (mean and maximum SUVs) will be determined over the prostate bed and over any acetate-avid or CT-identified suspicious lesions. The change in these SUVs with treatment will be assessed, as well as the number of lesions. A blinded second reviewer from Nuclear Medicine will reviewed all baseline and response PET-acetate scans.

SECONDARY OUTCOMES:
Prostate cancer response to treatment and progression (excluding PET Acetate assessment) | Time of enrollment up to two years
  Correlation with chemotherapy response

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Vaena, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No